CLINICAL TRIAL: NCT03784131
Title: Phase I Open-label, First-in-human Study to Evaluate Feasibility and Safety of Tissue Engineered Veins in Patients With Chronic Venous Insufficiency
Brief Title: Tissue Engineered Veins in Patients With Chronic Venous Insufficiency
Acronym: TECVI-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Verigraft AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-004021-13
Record Dates: First submitted 2018-11-16; First posted 2018-12-21 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Chronic Venous Insufficiency
Keywords: CVI; Leg Ulcer; Tissue Engineering; Personalized Vascular Graft; Chronic Venous Insufficiency; ATMP
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Tissue Engineered Vein (Experimental): P-TEV
  Interventions: Drug: P-TEV

INTERVENTIONS:
Drug: P-TEV — Replacement of vein with failing valves with personalized tissue engineering vein containing functional valves

SUMMARY:
This study aims to evaluate the safety (incidence of adverse events including serious adverse events and clinical significant laboratory abnormalities) of personalized tissue engineered veins (P-TEV) with valves implanted in patients with severe chronic venous insufficiency (CVI). For each patient a segment of the femoral vein containing the non-functioning valve will be surgically replaced with a single P-TEV containing a functioning valve.

DETAILED DESCRIPTION:
The advanced therapy medicinal product (ATMP) described herein is a personalized tissue- engineered vein (P-TEV) graft for use in surgical implantation to replace a defective or missing part of a patient's vein.

In this specific application a P-TEV graft with a functioning venous bicuspid valve is implanted to replace a nonfunctioning venous valve in the femoral vein of a patient suffering from severe CVI. The P-TEV graft for surgical implantation is 4-6 cm in length.

The P-TEV drug substance consists of an extracellular matrix (ECM) scaffold in the form of a decellularized (DC) allogeneic vein scaffold which is populated with autologous components from the patient's own peripheral whole blood (PWB) in an ATMP manufacturing process performed under GMP. As the allogeneic immunogenic material has been removed from the donated vein segment by DC and as the perfusion uses autologous PWB, no immunosuppression is required.

Successful implantation and treatment should prevent the reverse blood flow, decrease blood pooling in the lower leg, and thereby alleviate symptoms such as swelling, pain, and ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years (inclusive)
* CVI patients with painful swelling and/or skin changes and/or recurrent leg ulcer despite optimal conservative treatment for a period of time according to the investigator's judgement
* Patients with deep venous reflux (grade 3 and above)
* Meeting ASA (American Society of Anesthesiologists Classification) class 1 or 2 according to the PIs criteria
* Laboratory values

  * INR <1.7 (in case the patient uses Warfarin, the test might be repeated after the anticoagulant change)
  * Platelets ≥ 100 x 10 9 /L
  * Hemoglobin ≥ 100 g/L
  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * ASAT ≤ 2.5 × ULN
  * ALAT ≤ 2.5 × ULN
* Ability to understand the requirements of the study, give direct or representative written informed consent, and comply with the study procedures

Exclusion Criteria:

* Patients incapable to give direct or representative written informed consent
* Patients unlikely to cooperate fully in the study and/or with an anticipated poor compliance
* Non-walking patients or patients with lost ankle joint function
* Patients previously organ-transplanted
* Patients with cancer except in-situ stage cancer (basal-cell carcinomas and/or cervix cancer) and five year recurrence free period after treatment
* Patients with autoimmune diseases including rheumatoid arthritis, SLE and MS
* Pregnant or breast feeding women
* Patients with ongoing estrogen treatment for example for contraception. Alternative contraceptive methods (e.g. intrauterine device, bilateral tubal occlusion, vasectomized partner, sexual abstinence) should be used by women of reproductive age (defined as pre-menopausal female capable of becoming pregnant).
* BMI ≥ 35
* Patients who have participated in other clinical trials during the last 12 months
* Patients with artery pathology (ankle-brachial pressure index < 0,9 or > 1,3)
* Patients with thrombophilia according to the laboratory results at inclusion visit. One of the following criteria is needed for thrombophilia: Protein C < 40% or Protein S < 40 % or Leiden factor mutation or Antithrombin III < 40 % or present Lupus anticoagulant or Homocysteine > 1.5 ULN
* Patients with an active infection requiring systemic antibiotic treatment
* Patients with clinically significant cardiac disease (New York Heart Association, Class III or IV) or measured LVEF 40%
* Patients with uncontrolled hypertension
* Patients with renal dysfunction eGFR < 45 ml/min (according to the MDRD calculation)
* Patients with moderate or severe hepatic impairment (Child Pugh ≥ 7 points, i.e. class B or C)
* Patients with ongoing immunosuppression, systemic Cortisol treatment etc.
* Less than 3 months since previous ipsilateral venous intervention (e.g. Iliac recanalization)
* Clinically significant iliocaval stenosis or occlusion
* Current smoker of more than 20 cigarettes per day
* Other uncontrolled intercurrent illness that would jeopardize the patient's safety, interfere with the objectives of the protocol, or limit the patient's compliance with study requirements, as determined by the Investigator in consultation with the Sponsor
* Patients with severe SARSCoV-2 virus infection requiring hospitalization in the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Thrombosis leading to occlusion of the graft measured by Color Duplex Ultrasound | 12 months
  Ultrasonographic evaluation of occlusions of the graft.
Infection leading to surgical excision of the graft measured by blood samples | 12 months
  White blood cells count: >10 x10E9/L, C- Reactive Protein (CRP): >4 mg/L, sedimentation rate: >12mm).
Infection leading to surgical excision of the graft measured by Color Duplex Ultrasound | 12 months
  Ultrasonographic examination to assess infection of the graft
Infection leading to surgical excision of the graft measured by Computer Tomography | 12 months
  Infection of the graft assessed by Computer Tomography
Reporting of surgical complications | 12 months
  Perioperative surgical complications related to the implanted graft (technical failure leading to surgical failure).

SECONDARY OUTCOMES:
Change in symptoms assessed according to VCSS (Venous Clinical Severity Score) | 12 months
  The VCSS includes 9 hallmarks of venous disease, each scored on a severity scale from 0 (absent) to 3 (severe), plus a category for compression with higher scores representing greater compliance (still scale 0-3).
Change in symptoms assessed according to CEAP classification (clinical, etiologic, anatomic, pathophysiologic) | 12 months
  CEAP classification is assessed on scale from C0 (No visible or palpable signs of venous disease) to C6 (Active venous ulcer).
Health Related Quality of Life assessed by VEINES questionnaire | 12 months
  Responses are made on a 2- to 7-point scale that rates intensity, frequency, and agreement. Higher scores are associated with better quality-of-life.The focus of VEINES is on physical symptoms as opposed to psychological or social aspects.
Health Related Quality of Life assessed by EQ-5D-5L questionnaire | 12 months
  EQ-5D-5L is a standardized self-assessment instrument for health status.It has two components; health state description and evaluation.
  The first part contains 5 items with five levels of response regarding five dimensions (mobility, hygiene, activities, pain and anxiety).The five questions are compounded into a health index according to a mathematical formula validated against the population in several countries.The second part of the questionnaire comprises a standard vertical 20-cm VAS that is calibrated from 'the worst health you can imagine' (scored 0) at its base to 'the best health you can imagine' (scored 100) at its apex. Respondents are asked to 'mark an X on the scale to indicate how your health is TODAY' and to write the number in an adjoining box.
Durability of the P-TEV assessed by Color Duplex Ultrasound | 12 months
  The time period in which the valve contained in the implant retains its function verified by ultrasonographic examination.
Vessel dilatation in the implant assessed by Duplex Color Ultrasound | 12 months
  Ultrasonographic examination of vessel dilatation
Flow abnormalities in the implant assessed by Duplex Color Ultrasound | 12 months
  Ultrasonographic examination of flow abnormalities
Wall degeneration in the implant assessed by Duplex Color Ultrasound | 12 months
  Ultrasonographic examination of wall degeneration

CONTACTS AND LOCATIONS:
Overall Officials: Björquist, Study Director — Verigraft AB
Locations (1):
- Junta de Andalusia, Seville, Spain